CLINICAL TRIAL: NCT01555190
Title: Combination Therapy With Myo-inositol and Folic Acid Versus Myo-inositol Alone: Effects of Six Months Treatment on Clinical, Endocrine and Metabolic Features in Obese Women With Polycystic Ovary Syndrome
Brief Title: Combination Therapy With Myo-inositol and Folic Acid Versus Myo-inositol Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Maurizio Guido, medical doctor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000102012
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Polycystic Ovary Syndrome; Hirsutism; Menstrual Irregularity
Keywords: myo-inositol; folic acid
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hirsutism; Menstruation Disturbances | interventions — Folic Acid

ARMS (2):
- myo-inositol 1500 gr (Active Comparator): 6 months treatment with myo-inositol 1500 gr
  Interventions: Drug: myo-inositol 1500 gr
- myo-inositol 2000gr + folic acid 200 mcg (Active Comparator)
  Interventions: Drug: myo-inositol 2000 gr + folic acid 200 mcg

INTERVENTIONS:
Drug: myo-inositol 1500 gr
  Arms: myo-inositol 1500 gr
Drug: myo-inositol 2000 gr + folic acid 200 mcg
  Arms: myo-inositol 2000gr + folic acid 200 mcg

SUMMARY:
Previous studies have demonstrated that Myo-inositol is capable of restoring spontaneous ovarian activity, and consequently fertility, in most patients with PCOS. The aim of our study is to investigate the role of folic acid conteined in the inositol preparation. The study group included 50 patients, randomly allocated to subgroup A (myo-inositol 1500 gr) and subgroup B (myo-inositol 2000 gr + folic acid 200 mcg). The investigation include menstrual pattern and hirsutism score evaluation, hormonal assays, oral glucose tolerance test, euglycemic hyperinsulinaemic clamp and lipide profile at baseline and after six months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* women with PCOS diagnosed in accordance with Rotterdam Consensus Conference Criteria 2003
* BMI > 25 kg/m2
* age 18-35 years

Exclusion Criteria:

* pregnancy
* significant liver or renal impairment
* other hormonal dysfunctions (hypothalamic, pituitary, thyroidal or adrenal causes for the clinical signs)
* neoplasms
* unstable mental illness
* diagnosis of diabetes mellitus or impaired glucose tolerance
* use of drugs able to interfere with gluco-insulinaemic metabolism for at least three months prior entering the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
number of cycles in six months of therapy | 6 months
  We'll estimate the efficacy of the two treatments on the ovarian function and menstrual pattern.

SECONDARY OUTCOMES:
effects on oral glucose tollerance test | six months
effects on hoormonal assay | 6 months
effects oon lipide profile | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy